CLINICAL TRIAL: NCT06778772
Title: Transition to Adult Care in Epilepsy
Brief Title: Transition From Pediatric to Adult Epilepsy Care
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: tra epi
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy
Keywords: epilepsy; transition
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: transition pathway to adult care services for epilepsy patients. — This proposal aims to create a coordinated and shared transition pathway between pediatric and adult epilepsy services, addressing the needs of patients with chronic conditions. The primary objective is to assess the readiness of both patients and their caregivers for the transition, by comparing the Transition Readiness Assessment (TRAQ) questionnaire results between the last pediatric neuropsychiatric visit and the first adult neurology visit. Secondary objectives include evaluating changes in emotional-behavioral issues and quality of life, using the CBCL, YSR, and PedsQoL questionnaires. Assessments will be conducted at both pediatric and adult epilepsy services. The ultimate goal of the transition protocol is to improve care and outcomes for adolescents and young adults during the transition, focusing on emotional-behavioral and psychosocial aspects, and to develop a best-practice model that could influence future guidelines.

SUMMARY:
The goal of this observational study is to assess the preparation of the caregiver and the patient for the transition, by comparing the results of the Transition Readiness Assessment (TRAQ) questionnaire at the time of the last pediatric neuropsychiatric visit, which is then repeated at the first adult epilepsy neurology visit.

The assessments will be conducted at the last evaluation at the pediatric epilepsy service and repeated at the first visit to the adult epilepsy service.

DETAILED DESCRIPTION:
Epilepsy is a common pediatric neurological condition, with an incidence of 5-7 cases per 10,000 children and adolescents. In many cases, epilepsy does not remit in adulthood, requiring a transition from pediatric to adult epilepsy care. This transition should ideally be a planned and coordinated process addressing the patient's medical, psychosocial, and educational needs.

At the IRCCS C. Mondino Institute, around 700 pediatric epilepsy patients are followed, many with complex, genetically-based epilepsy and neuropsychiatric comorbidities. Transition programs, though essential, are challenging to implement, as pediatric and adult services often operate independently.

The transition period offers an opportunity for reassessment of care and the management of comorbidities, as well as counseling on aspects like education and independence. Psychiatric comorbidities can complicate the transition and negatively impact patients' quality of life. The Mondino Institute has developed a collaborative transition model involving both pediatric neuropsychiatrists and adult neurologists to address these challenges and better manage psychiatric comorbidities, ensuring a smoother transition to adult care.

The primary objective is to improve the multidisciplinary care of patients with epilepsy and psychiatric comorbidities, by implementing specific diagnostic and therapeutic evaluations for these comorbidities in patients transitioning from the pediatric and adolescent epilepsy center to the adult epilepsy service.

Secondary objectives include:

Defining the management pathway for psychiatric comorbidities in patients transitioning to adult epilepsy services, by identifying suitable structures and professionals for psychiatric and rehabilitative follow-up.

Optimizing the selection of specific pharmacological therapies for medium- to long-term maintenance.

In summary, the focus is on improving the care and treatment of epilepsy patients with psychiatric comorbidities, ensuring proper follow-up and therapeutic planning as they transition from pediatric to adult care.

ELIGIBILITY:
**Inclusion Criteria:**

* Patients aged 17 or 18 years.
* Diagnosed with focal or generalized epilepsy, regardless of etiology and neuropsychological, neuropsychiatric, or internal comorbidities.
* Those for whom continued epileptology follow-up is required according to standard care guidelines.

**Exclusion Criteria:**

* Patients undergoing EEG only for the detection of EEG abnormalities without a diagnosis of epilepsy.
* Patients for whom the last neuropsychiatric evaluation does not recommend continued epileptology follow-up (patients considered "cured" from epilepsy according to ILAE guidelines).

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patient with epilepsy primary care clinic
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
readiness for transition evaluated throughout Transition Readiness Assessment Questionnaire (TRAQ) | 1 year
  To evaluate the preparation of patients and caregivers for the transition process, the Transition Readiness Assessment Questionnaire (TRAQ) will be assessed, and scores will be compared across T0, T1, and T2.
  The TRAQ has a scale range from 0 to 5, where: 0 indicates insufficient readiness for transition; 5 indicates optimal readiness for transition.
  Higher scores indicate better preparation for the transition process, while lower scores suggest poorer readiness and a need for further support.

SECONDARY OUTCOMES:
to measure the efficacy of the transition process from pediatric to adult care using Transition Success in Childhood and Adolescence (TSCA) | 1 year
  To assess the efficacy of the completed transition protocol, the Transition Success in Childhood and Adolescence (TSCA) will be administred. TSCA scores will be compared across T0, T1, and T2.
  TSCA questionnaire has a scale range from 0 to 100, where: 0 represents the lowest level of transition success (poorest outcome), 100 represents the highest level of transition success (best outcome). Higher scores indicate a better outcome, reflecting greater success in the transition process, while lower scores indicate a poorer outcome and a need for further support.
To assess quality of life among patients and their families using Pediatric Quality of Life Inventory (PedsQL) | 1 year
  To explore perceptions of quality of life among patients and their families, Pediatric Quality of Life Inventory (PedsQL)scores will be analyzed across T0, T1, and T2. PedsQL has a scale range from 0 to 100, where: - 0 indicates the poorest quality of life, - 100 indicates the best possible quality of life. Higher scores reflect a better perception of quality of life, while lower scores suggest a lower quality of life and may indicate areas for improvement.
Behavioral and emotional issues will be evaluated by comparing the results of the Achenbach Child Behavior Checklist (ABCL) and Achenbach System of Empirically Based Assessment (ASR) | 1 year
  Behavioral and emotional issues will be evaluated by comparing the results of the Achenbach Child Behavior Checklist (ABCL) and Achenbach System of Empirically Based Assessment (ASR) between T0 and T2.
  ABCL is for children and adolescents (ages 1.5-18 years) and involves parent/caregiver reports.
  ASR is for adolescents (12-18) and adults (18+), and it can be used as a self-report or informant report tool.
  Scores for both measures typically range from 0 to 3. 0 indicates no problem, 3 indicates a severe problem. Higher scores indicate more significant behavioral or emotional issues, while lower scores suggest fewer or no problems.
To understand the factors influencing transition readiness and to identify potential barriers, the Transition NEEDS Questionnaire will be developed. | 1 year
  To provide a comprehensive understanding of the factors influencing transition readiness and to identify potential barriers, the Transition NEEDS Questionnaire will be developed. This semi-structured, qualitative interview for clinicians systematically assesses six critical domains: patient and family readiness, diagnostic gaps, therapeutic gaps, social/care support gaps, educational/work-related gaps, psychological/emotional gaps. This tool, grounded in clinical and theoretical literature, offers a systematic and practical method for evaluating the complex needs of patients transitioning from pediatric to adult epilepsy care.
To assess the qualitative aspects of the transition phase througout a qualitative scale | 1 year
  The TRANS-EPI Questionnaire focuses on qualitative aspects of the transition phase, exploring: timing and introduction to the transition process; evaluation of information proovided; expectations from adult neurology care; concerns about continuity of care and autonomy

CONTACTS AND LOCATIONS:
Overall Officials: Valentina De Giorgis, MD, Principal Investigator — Child and Adolescent Epileptology
Locations (1):
- Child Neuropsichiatry, Pavia, Italy

REFERENCES:
- [Background] Andrade DM, Bassett AS, Bercovici E, Borlot F, Bui E, Camfield P, Clozza GQ, Cohen E, Gofine T, Graves L, Greenaway J, Guttman B, Guttman-Slater M, Hassan A, Henze M, Kaufman M, Lawless B, Lee H, Lindzon L, Lomax LB, McAndrews MP, Menna-Dack D, Minassian BA, Mulligan J, Nabbout R, Nejm T, Secco M, Sellers L, Shapiro M, Slegr M, Smith R, Szatmari P, Tao L, Vogt A, Whiting S, Carter Snead O 3rd. Epilepsy: Transition from pediatric to adult care. Recommendations of the Ontario epilepsy implementation task force. Epilepsia. 2017 Sep;58(9):1502-1517. doi: 10.1111/epi.13832. Epub 2017 Jul 6. PMID 28681381
- [Background] Borlot F, Tellez-Zenteno JF, Allen A, Ali A, Snead OC 3rd, Andrade DM. Epilepsy transition: challenges of caring for adults with childhood-onset seizures. Epilepsia. 2014 Oct;55(10):1659-66. doi: 10.1111/epi.12752. Epub 2014 Aug 28. PMID 25169716